CLINICAL TRIAL: NCT05488951
Title: The Effects of strEngth aNd BaLance Exercise on Executive Function in People Living With Dementia (ENABLED): A Randomized Controlled Trial
Brief Title: The Influence of the Otago Exercise Program on Executive Function Among People Living With Mild to Moderate Dementia
Acronym: ENABLED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Deborah Jehu, Assistant Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1838020
Record Dates: First submitted 2022-07-28; First posted 2022-08-05 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Dementia
Keywords: Dementia; Otago Exercise Program; Executive Function
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: For this pilot study, participants will be randomly assigned (1:1) to the exercise (n=21) or control group (n=21). The statisticians (Dr Jennifer Waller and Dr. Brittany Ange) will generate the randomization sequence and provide it to the study coordinator after the baseline assessment; they will also conceal the treatment allocation from the assessors. Randomization will be stratified by biological sex (female/male) and study site. Blocked randomization will be performed using random block sizes of 2 and 4. Permutations of exercise or control will be performed in each block.
Who Masked: Outcomes Assessor
Masking Description: The investigators conducting the testing will be masked to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago Exercise Program Plus Usual Care (Experimental): The Otago Exercise Program will be led by a physical therapist in a group setting (5-7 participants/exercise class). The exercise will be 20 min of walking and 30 min of strength and balance exercises 3x/week for 6 months. The physical therapist will select suitable exercises for each participant, such that the exercise is individualized and progressive. Participants will also receive usual care from health care providers (e.g., specialist and local doctor visits, community nurse visits, paid care provider visits, hospitalizations as required, and any ongoing treatment for any illness and/or their comorbidities).
  Interventions: Other: Otago Exercise Program
- Usual Care Only (No Intervention): Usual care will consist of routine care from their health care providers (e.g., specialist and local doctor visits, community nurse visits, paid care provider visits, hospitalizations as required, and any ongoing treatment for any illness and/or their comorbidities).

INTERVENTIONS:
Other: Otago Exercise Program — The Otago Exercise Program will be led by a physical therapist in a group setting (5-7 participants/exercise class). The exercise will be 20 min of walking and 30 min of strength and balance exercises (i.e., 50 min exercise class) 3x/week for 6 months. The physical therapist will select suitable exercises for each participant, such that the exercise is individualized and progressive.
  Arms: Otago Exercise Program Plus Usual Care

SUMMARY:
The primary aim of this study is to conduct a pilot 6-month assessor-blinded randomized controlled trial to determine if the Otago Exercise Program plus usual care improves executive function in people living with mild to moderate dementia compared to usual care among those living in a nursing home or assisted living facility. The exploratory aims are to determine if the Otago Exercise Program plus usual care improves inflammatory blood biomarkers, kynurenine metabolites, epigenetics, mobility, balance, cognition, mood, fall-related self-efficacy, health-related quality of life, sleep, physical activity, and falls by sex and race compared to usual care alone among people living with mild to moderate dementia.

DETAILED DESCRIPTION:
Dementia is a growing public health problem. Approximately 46.8 million individuals worldwide were living with dementia in 2015, which is estimated to reach 131.5 million by 2050. The global healthcare expenditure of dementia was $604 billion in 2010, which is projected to dramatically increase. Therefore, there is an urgent need to alleviate this growing public health concern.

Executive function is important for maintaining independence in activities of daily living; yet, people living with dementia often have poor executive function. Executive function includes the abilities to: make decisions, reason, problem-solve, initiate and maintain tasks, as well as adapt to changing cognitive conditions. Poor executive function is linked with other important health markers, such as poor physical function, falls, and mortality. It is possible that these poor health outcomes in people living with dementia may, in part, be explained by shared mechanisms including inflammation, autophagy, and apoptosis. Interestingly, these poor health outcomes among people living with dementia seem to depend on sex and race, with females and African Americans exhibiting greater comorbidities; nevertheless, the underlying mechanisms are poorly understood.

Poor executive function is linked with other important health markers, such as poor physical function and falls via reduced judgement and self-regulation. Cognitive and physical frailty are frequently observed together, likely due to common pathophysiological mechanisms. People living with dementia are often frail and prone to multiple tipping point incidents, potentially leading to adverse health outcomes. Cognitive and physical frailty also seems to depend on sex and race, with females and African Americans exhibiting a higher incidence of dementia; nevertheless, the underlying mechanisms are poorly understood. Overall, people living with dementia often have multiple comorbidities and complex medical needs; thus, research targeted at addressing these health disparities should be a frontline priority.

Exercise may be a viable strategy to improve executive function in people living with dementia. Mounting evidence suggests that strength and balance interventions (≥3x/week) are safe and effective at improving cognition and mobility, as well as reducing falls in cognitively intact community-dwelling older adults. Yet, historically, people living with dementia have been systematically excluded from intervention studies due to researchers' ineligibility criteria. Few studies have examined the influence of exercise on executive functioning among people living with dementia, but have shown no effect; it is possible that the small sample sizes may have contributed to these null findings. Therefore, further research is warranted to improve executive function and other health outcomes among people living with mild to moderate dementia.

ELIGIBILITY:
Inclusion criteria

* Aged 55 years and older
* Reside in a nursing home or assisted living facility
* Have any type of mild to moderate dementia confirmed by medical records and/or a physician
* Can read, write, and speak English with acceptable visual and auditory acuity
* Able to walk 3 meters with or without the assistance of another person
* Have a legally authorized representative who can provide informed consent
* Able to provide assent
* Able to understand and follow instructions
* Have a life expectancy of ≥12 months as estimated by a healthcare provider

Exclusion criteria

* Reside in the community
* Severe dementia (e.g., Montreal Cognitive Assessment ≤6/30) and are not able to follow instructions
* Severe psychiatric condition
* Progressive neurological disease other than dementia (i.e., neurological disease, such as Parkinson's, that is mild and stable is not an exclusion)
* Delirium
* Acute medical condition
* Medical condition precluding exercise (e.g., unstable cardiac disease)
* Recent surgery affecting mobility
* Enrolled in another research study
* Blindness
* Aphasia
* Enrolled in another research study
* Receiving hospice care

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Color Word Stroop Test | Baseline, 6 months
  Response inhibition involves deliberately suppressing dominant, automatic, or prepotent responses, and will be assessed using the Stroop Colour-Word Test. For the Stroop Test, there will be three conditions. First, participants will be asked to read aloud words printed in black ink (e.g., BLUE). Second, they were instructed to read aloud the color of colored rectangles. Finally, they will shown a page of color-words printed in incongruent colored ink (e.g., the word "BLUE" printed in red ink). Participants will be asked to name the ink color in which the words are printed (while ignoring the word itself). There will 50 trials for each condition and the time taken to read each condition will recorded.

SECONDARY OUTCOMES:
Change in the Digit Symbol Substitution Test | Baseline, 6 months
  The Digit Symbol Substitution Test is a measure of processing speed and consists of nine digit-symbol pairs. Participants will be asked to fill in as many corresponding symbols for the given digits within 90 s, with a greater number of items correctly coded indicating better processing speed. Performance will be measured by the number of correct symbols; a greater number of symbols indicates better performance.
Change in the oral Trail Making Test | Baseline, 6 months
  Set-shifting will be assessed using the oral Trail-Making Test Part B minus A. It will involve going back and forth between multiple tasks or mental sets. Part A will assess psychomotor speed; participants will count numbers aloud in sequential order, starting at 1 and ending at 25. We will record the amount of time (in seconds) for the participants to complete the task. Part B will consist of orally switching back and forth from numbers to letters (the numbers extend from 1 to 13 and the letters from A to L). Participants will be instructed to orally count as quickly and as accurately as possible from 1 to A, A to 2, 2 to B, B to 3, and so on, until they complete the task. We will record the amount of time (in seconds) for participants to complete the task. To index set shifting, the completion time difference between Part B and Part A will be calculated. Smaller difference scores indicate better set shifting.
Change in the Digit Span Forwards and Backwards | Baseline, 6 months
  Working memory will be assessed using the verbal digit span forward and backward task. This task involves presenting a series of random digits (from 1 to 9), after which participants will be asked to verbally repeat the list in the same order and in the reverse order, respectively, in separate trials. If successful, they will be provided a longer number sequence. The total number of correct trials and the longest correct trial will be recorded.
Change in the Rey Auditory Verbal Learning Test | Baseline, 6 months
  The Rey Auditory Verbal Learning Test is a measure of learning and short-term memory. We will read a list of 15 words and participants will be asked to recall as many words as they can remember. We will record the total recall, intrusions, and repetitions for: immediate recall, delayed recall, and word recognition.
Change in the Benton Judgement of Line Orientation | Baseline, 6 months
  Perception will be assessed using the Benton Judgement of Line Orientation. Participants will be presented with 15 pairs of lines. Participants will judge the angle of both lines with respect to the reference line angle. The total score ranges from 0 to 15.
Change in the Boston Naming Test | Baseline, 6 months
  Language skills will be assessed with the Boston Naming Test, which involves visually looking at 15 printed pictures on a piece of paper and verbalizing the name of the objects. The total score ranges from 0 to 15.
Change in Health Utilities Index-3 | Baseline, 6 months
  The Health Utilities Index-3 is a questionnaire related to quality of life. We will use the total score as the outcome measure.
Change in the Visual Analogue Scale | Baseline, 6 months
  The Visual Analogue Scale (VAS) is a measure of overall perceived rating of health. The endpoint of 100 is labelled "The best health you can imagine" while a score of 0 was labelled "The worse health you can imagine". Participants will be asked to report their perceived health on the day of the assessment.
Change in the Geriatric Depression Scale | Baseline, 6 months
  The Geriatric Depression Scale is a 15-item questionnaire that assesses depressed mood. A score of greater than 5 points is suggestive of depression, while a score of greater than or equal to a score of 10 is almost always indicative of depression.
Change in the short-Falls Efficacy Scale International | Baseline, 6 months
  The Short-Falls Efficacy Scale International measures fear when performing 7 daily activities. Scores between 7-8 are indicative of low concern for falling, 9-13 are indicative of moderate concern for falling, and 14-28 are indicative of high concern for falling.
Change in Functional Comorbidity Index | Baseline, 6 months
  The Functional Comorbidity Index includes 18 evenly weighted comorbidities that stratify on physical functional status. This scale's score was the total number of comorbidities.
Change in body composition (weight (kg)) | Baseline, 6 months
  Change in body composition will be measured using the Omron Body Composition Monitor. We will record weight (kg).
Change in body composition (fat (%)) | Baseline, 6 months
  Change in body composition will be measured using the Omron Body Composition Monitor. We will record body fat composition (%).
Change in body composition (muscle (%)) | Baseline, 6 months
  Change in body composition will be measured using the Omron Body Composition Monitor. We will record skeletal muscle composition (%).
Change in the Short Physical Performance Battery | Baseline, 6 months
  The Short Physical Performance Battery is a valid and reliable measure of physical performance and is comprised of three components, including: balance, gait, and chair stands. Balance will be assessed over 10 s of stance with feet together, semi-tandem, and tandem stance. Gait speed will be measured over 4 m with a stopwatch. The five times sit to stand will be measured with a stopwatch. The total score ranges from 0 worst) to 12 (best).
Change in dual-task posture (sway area (degrees/s squared)) | Baseline, 6 months
  Dual-task posture will be measured with APDM inertial sensors. Dual-task posture will involve standing with feet apart with no cognitive task, as well as while counting backwards by 1's. We will examine sway area (degrees/s squared).
Change in dual-task posture (root mean square sway (degrees)) | Baseline, 6 months
  Dual-task posture will be measured with APDM inertial sensors. Dual-task posture will involve standing with feet apart with no cognitive task, as well as while counting backwards by 1's. We will examine root mean square sway (degrees).
Change in dual-task posture (frequency of sway (Hz)) | Baseline, 6 months
  Dual-task posture will be measured with APDM inertial sensors. Dual-task posture will involve standing with feet apart with no cognitive task, as well as while counting backwards by 1's. We will examine frequency of sway (Hz).
Change in dual-task posture (jerk (m²/s^5)) | Baseline, 6 months
  Dual-task posture will be measured with APDM inertial sensors. Dual-task posture will involve standing with feet apart with no cognitive task, as well as while counting backwards by 1's. We will examine jerk (m²/s^5).
Change in dual-task posture (mean velocity (m/s)) | Baseline, 6 months
  Dual-task posture will be measured with APDM inertial sensors. Dual-task posture will involve standing with feet apart with no cognitive task, as well as while counting backwards by 1's. We will examine mean velocity (m/s)
Change in dual-task posture (path length(m/s²)) | Baseline, 6 months
  Dual-task posture will be measured with APDM inertial sensors. Dual-task posture will involve standing with feet apart with no cognitive task, as well as while counting backwards by 1's. We will examine path length(m/s²).
Change in dual-task gait (gait speed (m/s)) | Baseline, 6 months
  Dual-task gait will be measured with APDM inertial sensors. Dual-task gait will involve walking 4 m with no cognitive task as well as while naming all the words starting with a specific letter. We will examine gait speed (m/s).
Change in dual-task gait (double support (%)) | Baseline, 6 months
  Dual-task gait will be measured with APDM inertial sensors. Dual-task gait will involve walking 4 m with no cognitive task as well as while naming all the words starting with a specific letter. We will examine double support (%).
Change in dual-task gait (stride length (m)) | Baseline, 6 months
  Dual-task gait will be measured with APDM inertial sensors. Dual-task gait will involve walking 4 m with no cognitive task as well as while naming all the words starting with a specific letter. We will examine stride length (m).
Change in dual-task gait (upper body range of motion (degrees)) | Baseline, 6 months
  Dual-task gait will be measured with APDM inertial sensors. Dual-task gait will involve walking 4 m with no cognitive task as well as while naming all the words starting with a specific letter. We will examine upper body range of motion (degrees).
Change in dual-task mobility (task duration (s)) | Baseline, 6 months
  Dual-task mobility will be assessed with the timed-up-and-go (TUG). The TUG involves getting up from a chair, walking 3 m, turning around, walking back, and sitting down. Participants will complete the TUG with no cognitive task, as well as while completing a category task. We will examine task duration (s).
Change in dual-task mobility (turn duration (s)) | Baseline, 6 months
  Dual-task mobility will be assessed with the timed-up-and-go (TUG). The TUG involves getting up from a chair, walking 3 m, turning around, walking back, and sitting down. Participants will complete the TUG with no cognitive task, as well as while completing a category task. We will examine turn duration (s).
Change in dual-task mobility (turn velocity (degrees/s)) | Baseline, 6 months
  Dual-task mobility will be assessed with the timed-up-and-go (TUG). The TUG involves getting up from a chair, walking 3 m, turning around, walking back, and sitting down. Participants will complete the TUG with no cognitive task, as well as while completing a category task. We will examine turn velocity (degrees/s).
Change in dual-task mobility (lean angle (degrees)) | Baseline, 6 months
  Dual-task mobility will be assessed with the timed-up-and-go (TUG). The TUG involves getting up from a chair, walking 3 m, turning around, walking back, and sitting down. Participants will complete the TUG with no cognitive task, as well as while completing a category task. We will examine lean angle (degrees).
Change in turning (task duration (s)) | Baseline, 6 months
  Turning will be assessed with a 360 degree turn with APDM inertial sensors. We will examine task duration (s).
Change in turning (turn angle (degrees)) | Baseline, 6 months
  Turning will be assessed with a 360 degree turn with APDM inertial sensors. We will examine turn angle (degrees).
Change in turning (turn velocity (degrees/s)) | Baseline, 6 months
  Turning will be assessed with a 360 degree turn with APDM inertial sensors. We will examine turn velocity (degrees/s).
Change in functional lower extremity strength (task duration (s)) | Baseline, 6 months
  Functional lower extremity strength will be assessed with the five times sit to stand using APDM inertial sensors. We will examine task duration (s).
Change in functional lower extremity strength (lean angle (degrees)) | Baseline, 6 months
  Functional lower extremity strength will be assessed with the five times sit to stand using APDM inertial sensors. We will examine lean angle (degrees).
Change in hand grip strength | Baseline, 6 months
  To measure hand grip strength, participants will be asked to hold the dynamometer in their hand, with the arm parallel to the side of the body. Participants will then squeeze the dynamometer with maximum isometric effort for about 3-5 seconds. The average of two trials will be recorded for the right and left hands.
Change in quadriceps grip strength | Baseline, 6 months
  We will use the JTECH Commander handheld dynamometer to measure quadriceps strength. From the seated position, the investigator will secure a strap around the participants' lower shank and a secured object, such that the lower shank is at 60 degrees from flexion. Participants will extend their knee with maximum isometric effort for about 3-5 seconds. The average of two trials will be recorded for the right and left legs.
Change in physical activity (% of time in different levels of physical activity) | Baseline, 6 months
  An Axivity Monitor will be worn on the wrist over 7 days and will measure physical activity. The Axivity Monitor will provide information: percentage of time in light, moderate, vigorous, and very vigorous activity (%).
Change in physical activity (step count) | Baseline, 6 months
  An Axivity Monitor will be worn on the wrist over 7 days and will measure physical activity. The Axivity Monitor will provide information: average daily step count (steps).
Change in physical activity (number of sedentary bouts) | Baseline, 6 months
  An Axivity Monitor will be worn on the wrist over 7 days and will measure physical activity. The Axivity Monitor will provide information: number of sedentary bouts (count).
Change in physical activity (time in sedentary bouts (min)) | Baseline, 6 months
  An Axivity Monitor will be worn on the wrist over 7 days and will measure physical activity. The Axivity Monitor will provide information: average time in sedentary bouts (min).
Change in sleep efficiency (total sleep time/total time in bed) | Baseline, 6 months
  An Axivity Monitor will be worn on the wrist over 7 days and will measure sleep. The Axivity Monitor will provide information: sleep efficiency (total sleep time/total time in bed).
Change in sleep (number of awakenings) | Baseline, 6 months
  An Axivity Monitor will be worn on the wrist over 7 days and will measure sleep. The Axivity Monitor will provide information: number of awakenings (number).
Change in sleep (average awake length (min)) | Baseline, 6 months
  An Axivity Monitor will be worn on the wrist over 7 days and will measure sleep. The Axivity Monitor will provide information: average awake length (min).
Change in sleep (Sleep Fragmentation Index) | Baseline, 6 months
  An Axivity Monitor will be worn on the wrist over 7 days and will measure sleep. The Axivity Monitor will provide information: sleep fragmentation index. The Sleep Fragmentation Index = the sum of the Movement Index and Fragmentation Index. The Movement Index = the total of scored awake minutes divided by Total time in bed in hours x 100. The Fragmentation Index = the percentage of one-minute periods of sleep vs. all periods of sleep in the sleep period.
Falls | Retrospective and Prospective for 6 months
  Falls will be recorded by the nursing home or assisted living facility staff on incident reports.
Change in inflammatory blood biomarkers (Interleukin-6) | Baseline, 6 months
  We will draw blood at baseline and 6 months. We will examine inflammatory blood biomarkers, including Interleukin-6 (ng/ml), measured using multiplex assay.
Change in inflammatory blood biomarkers (Interleukin-1) | Baseline, 6 months
  We will draw blood at baseline and 6 months. We will examine inflammatory blood biomarkers, including Interleukin-1α (ng/µg), measured using multiplex assay.
Change in inflammatory blood biomarkers (Tumor Necrosis Factor-α) | Baseline, 6 months
  We will draw blood at baseline and 6 months. We will examine inflammatory blood biomarkers, including Tumor Necrosis Factor-α (ng/ml), measured using multiplex assay.
Change in kynurenine pathway metabolites (kynurenine) | Baseline, 6 months
  We will draw blood at baseline and 6 months. We will examine kynurenine pathway metabolites, including kynurenine (ng/ml), measured using mass spectroscopy.
Change in kynurenine pathway metabolites (tryptophan) | Baseline, 6 months
  We will draw blood at baseline and 6 months. We will examine kynurenine pathway metabolites, including tryptophan (µmol/L), measured using mass spectroscopy.
Change in kynurenine pathway metabolites (kynurenic acid) | Baseline, 6 months
  We will draw blood at baseline and 6 months. We will examine kynurenine pathway metabolites, including kynurenic acid (ng/ml), measured using mass spectroscopy.
Change in epigenetics | Baseline, 6 months
  We will draw blood at baseline and 6 months. We will examine epigenetics (genome-wide test, global methylation, and aging clock). DNA samples will be extracted with Applied Biosystem MagMAX DNA Multi-Sample Ultra 2.0 kit using KingFisher Duo Prime automated system, quantified by NanoDrop 2000 Spectrophotometer system. Genome-wide DNA methylation analysis will be conducted using the Illumina Infinium MethylationEPIC BeadChip (Illumina Inc., Denver, CO) in DNA samples. DNA methylation beta values will be used to estimate the DNA methylation age (DNAm age) prior to normalization using the online epigenetic age calculator (http://dnamage.genetics.ucla.edu).

OTHER OUTCOMES:
Montreal Cognitive Assessment | Baseline
  The Montreal Cognitive Assessment (MOCA) is a measure of global cognition and is a screening tool for cognitive impairment. The MoCA also measures executive function, short-term memory recall, visuospatial abilities, attention, concentration and working memory, language, as well as orientation to time and place.
Morse Fall Scale | Baseline
  The Morse Fall Scale is a 6-item measure of fall-risk. The items in the scale are comprised of the history of falling, secondary diagnosis, ambulatory aids, intravenous therapy, gait, and mental status. A Morse Fall Scale score of 0-24 indicates no risk, 25-30 indicates low risk, and >=51 indicates high risk.
Cornell Depression Scale | Baseline
  The Cornell Depression Scale is a 19-item questionnaire that assesses depressed mood, and is examined by a clinician. A score of greater than 10 points is suggestive of probable major depression, while a score of greater than 18 points is suggestive of definite major depression.
Adverse Events | Monthly for 6 months
  Adverse events will be recorded by the nursing home or assisted living facility staff on incident reports.
Exercise adherence, measured by the average number of exercise sessions attended | 3x/week for 6 months
  Exercise adherence will be tracked at each exercise session in a logbook by a research assistant for each participant in the exercise program.
Intervention Satisfaction, measured on a Likert scale | 6 months
  The Otago Exercise Program plus usual care group will complete a questionnaire related to the exercise program satisfaction, which will be scored on a 1 (very unsatisfied) to 5 (very satisfied) scale. This questionnaire will only be given once to participants receiving the Otago Exercise Program at the end of their program.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Jehu, PhD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No